CLINICAL TRIAL: NCT02386683
Title: Intraoperative Lung-Protective Ventilation in Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, attending doctor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: kY2014-031-02
Record Dates: First submitted 2014-10-18; First posted 2015-03-12 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Ventilator-induced Lung Injury
Keywords: Protective mechanical ventilation; ventilator-induced lung injury; neurosurgery
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group L (Active Comparator): lung-protective ventilation applied in anesthesia
  Interventions: Other: lung-protective ventilation
- Group T (No Intervention): traditional ventilation applied in anesthesia

INTERVENTIONS:
Other: lung-protective ventilation — mechanical ventilated with a tidal volume of 6-8ml/kg ideal body weight (IBW) and 6-8 cm H2O PEEP in anesthesia
  Arms: Group L

SUMMARY:
The purpose of this study is to explore the effectiveness of lung-protective ventilation during general anesthesia for neurosurgical procedures on postoperative pulmonary outcome, compared with traditional ventilation.

DETAILED DESCRIPTION:
After screened for preoperative risk classification of postoperative respiratory complications,360 patients undergoing elective neurosurgery are randomly assigned to two groups, lung-protective ventilation (L) and traditional ventilation(T).Patients are mechanical ventilated with either a tidal volume of 10-12 ml/kg ideal body weight (IBW,T) or 6-8ml/kg IBW with 6-8 cm H2O PEEP(L),both with recruitment maneuver (RM).Each RM consists of applying a continuous positive airway pressure of 30 cmH2O for 30 seconds. Postoperative pulmonary complications are compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. > 40 years ,and < 80 years
2. Scheduled for neurosurgery
3. After informed consent has been obtained
4. With an expected duration of ≥ 4 hours
5. preoperative risk index for pulmonary complications≥ 2
6. Glasgow Coma Scale >8

Exclusion Criteria:

1. Mechanical ventilation of > 1 hour within the last 2 weeks before surgery
2. Body mass index ≥ 35 kg/m2
3. Acute respiratory failure (pneumonia, acute lung injury or acute respiratory distress syndrome)
4. Emergency surgery
5. Severe cardiac disease
6. Progressive neuromuscular illness
7. Pregnancy
8. Refusal to participate

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | 7 days after surgery
  modified Clinical Pulmonary Infection Score (mCPIS):Temperature,Blood leukocytes,Tracheal secretions,Oxygenation Pao2/Fio2,Chest radiograph; Grade scale for postoperative pulmonary complications:Grade 0 representing the absence of any pulmonary complication and grades 1 through 4 representing successively the worse forms of complications

SECONDARY OUTCOMES:
Intraoperative brain relaxation. | 1 day undergonging surgery
  using a four-point scale: 1, completely relaxed; 2, satisfactorily relaxed; 3, firm brain; 4, bulging brain;
The postoperative complications within 30 days | 30 days after surgery
  Surgical complications，Systematic complications; Septic shock， Death
Postoperative hypoxemia | 7 days after surgery
  PaO2 less than 60 mmHg, SpO2 less than 90%; PaO2 /FiO2 less than 300.
Peripheral blood inflammatory response indicators | 1 day after surgery
  interleukin 6, tumor necrosis factor TNF-α.
Postoperative antibiotic usage | 30 days after surgery
  antibiotic dose
Postoperative pulmonary complications | 30 days after surgery
  modified Clinical Pulmonary Infection Score (mCPIS):Temperature,Blood leukocytes,Tracheal secretions,Oxygenation Pao2/Fio2,Chest radiograph; Grade scale for postoperative pulmonary complications:Grade 0 representing the absence of any pulmonary complication and grades 1 through 4 representing successively the worse forms of complications
Unanticipated ICU treatment. | 30 days after surgery
  Unanticipated ICU treatment.
ICU stay and length of hospital stay | 30 days after surgery
  ICU stay and length of hospital stay
All cause of mortality at 30 days | 30 days after surgery
  mortality
Cost analysis | 30 days after surgery
  Data of total non-operative costs, costs per day.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, MD, Study Chair — Department of Anesthesiology, Beijing Tiantan Hospital， Capital Medical University; liyong Zhang, MD, Study Director — Department of Anesthesiology, Beijing Tiantan Hospital， Capital Medical University
Locations (1):
- Department of Anesthesiology,Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Xiong W, Peng Y, Zhang W, Han R. The effect of an intraoperative, lung-protective ventilation strategy in neurosurgical patients undergoing craniotomy: study protocol for a randomized controlled trial. Trials. 2018 Feb 2;19(1):85. doi: 10.1186/s13063-018-2447-4. PMID 29394907